CLINICAL TRIAL: NCT04896307
Title: The Impact of Organizational Leadership on Physician Burnout and Satisfaction at The Ottawa Hospital
Brief Title: The Impact of Organizational Leadership on Physician Burnout and Satisfaction
Status: Completed | Type: Observational
Sponsor: University of Ottawa (Other)
Collaborators: The Ottawa Hospital (Other); The Ottawa Hospital Research Institute (Unknown)
Responsible Party: Principal Investigator, Edward Spilg, Assistant Professor, University of Ottawa
Other Study IDs: 20200431-01H
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Burnout, Professional; Satisfaction; Leadership
Keywords: burnout; satisfaction; organizational leadership; survey
MeSH Terms: conditions — Burnout, Professional; Personal Satisfaction; Burnout, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians at The Ottawa Hospital: Online survey completed by physicians working at The Ottawa Hospital consisting of the 2-item Maslach Burnout Inventory, a Satisfaction Questionnaire and the 12-Item Participatory Management Leadership Score.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
Physician burnout is a global issue characterized by emotional exhaustion, depersonalization, and low levels of personal accomplishment. Recent evidence suggests that organization-directed interventions were more likely to lead to reductions in burnout when compared to physician-directed interventions. More specifically, the leadership behaviors of the direct physician supervisor play a critical role in the well-being of physicians they supervise.

As such, the aims of this project are: 1) To improve our understanding of the prevalence of burnout and professional satisfaction of physicians working at the Ottawa Hospital (TOH), and 2) To evaluate the relationship between the leadership qualities of direct physician supervisors (i.e. Division and Department Heads) and the well-being and burnout of their physicians. Specifically, a cross-sectional survey will be completed by physicians at TOH to assess their levels of burnout and satisfaction and the leadership qualities of their direct physician supervisors.

DETAILED DESCRIPTION:
Physician burnout is a global issue characterized by emotional exhaustion, depersonalization, and low levels of personal accomplishment. Burnout symptoms as high as 50% have been documented worldwide. According to the 2018 National Physician Health Survey, 30% of Canadian Physicians and Residents are experiencing burnout, with 26% high emotional exhaustion and 15% high depersonalization. Physician burnout is associated with low job satisfaction, decreased quality of patient care, reduced productivity, high job turnover, and early retirement from clinical practice. However, evidence suggests burnout is reversible and even preventable.

Recent evidence suggests that organization-directed interventions were more likely to lead to reductions in burnout when compared to physician-directed interventions. More specifically, the leadership behaviors of the direct physician supervisor play a critical role in the well-being of physicians they supervise. To date, we are unaware of any study that has examined the relationship between organizational leadership and degree of burnout and professional satisfaction in a Canadian tertiary care centre. Understanding physician burnout and professional satisfaction has strategic importance to the health of the physician, the patient, and the organization.

A recent study of 2813 physicians at the Mayo clinic found that each 1-point increase in supervisor's leadership score was associated with a 3.3% decrease in the likelihood of burnout and 9% increase in satisfaction of physicians. Furthermore, 11% and 47% of the variation of burnout and satisfaction, respectively, was attributed to the leadership rating of the physician's supervisor. The findings from this study further highlight the importance of prioritizing leadership as a key performance indicator, but it is necessary to first determine whether the Mayo Clinic's findings can be translated to a Canadian tertiary care centre.

As such, the aims of this project are: 1) To improve our understanding of the prevalence of burnout and professional satisfaction of physicians working at TOH, and 2) To evaluate the relationship between the leadership qualities of direct physician supervisors (i.e. Division and Department Heads) and the well-being and burnout of their physicians.

Our study will use Shanafelt et al's study as a guide to investigate leadership qualities at TOH. A cross-sectional online survey will be completed by physicians at TOH that will assess their levels of burnout and satisfaction and the leadership qualities of their direct physician supervisor.

ELIGIBILITY:
Inclusion Criteria:

* all physicians working at The Ottawa Hospital

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All physicians working at The Ottawa Hospital
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
2-item Maslach Burnout Inventory (MBI) | Baseline
  Burnout will be assessed by the 2-item version of the MBI.
Satisfaction Questionnaire | Baseline
  Overall satisfaction with TOH as a health care organization will be evaluated with the following question, rated on a 5-point Likert scale from "very satisfied" to "very dissatisfied": "Considering everything, how would you rate your overall satisfaction with TOH as a whole at the present time?"
12-Item Participatory Management Leadership Index | Baseline
  This validated questionnaire assesses the opinion of the leadership qualities of the physician's immediate supervisor. The 12 items assess specific characteristics of leadership that are measurable and actionable. Participants will also be asked to rate their overall satisfaction with their immediate supervisor on a 5-point Likert scale from "very satisfied" to "very dissatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Edward Spilg, MBChB, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maslach C, Jackson SE, Leiter MP. Maslach burnout inventory manual. Vol 4: Consulting psychologists press Palo Alto, CA; 1996.
- [Background] Linzer M, Visser MR, Oort FJ, Smets EM, McMurray JE, de Haes HC; Society of General Internal Medicine (SGIM) Career Satisfaction Study Group (CSSG). Predicting and preventing physician burnout: results from the United States and the Netherlands. Am J Med. 2001 Aug;111(2):170-5. doi: 10.1016/s0002-9343(01)00814-2. No abstract available. PMID 11498074
- [Background] Schaufeli WB, Leiter MP, Maslach C. Burnout: 35 years of research and practice. Career development international. 2009;14(3):204-220.
- [Background] Klein J, Grosse Frie K, Blum K, von dem Knesebeck O. Burnout and perceived quality of care among German clinicians in surgery. Int J Qual Health Care. 2010 Dec;22(6):525-30. doi: 10.1093/intqhc/mzq056. Epub 2010 Oct 8. PMID 20935011
- [Background] Panagopoulou E, Montgomery A, Benos A. Burnout in internal medicine physicians: Differences between residents and specialists. Eur J Intern Med. 2006 May;17(3):195-200. doi: 10.1016/j.ejim.2005.11.013. PMID 16618453
- [Background] Arigoni F, Bovier PA, Sappino AP. Trend of burnout among Swiss doctors. Swiss Med Wkly. 2010 Aug 9;140:w13070. doi: 10.4414/smw.2010.13070. eCollection 2010. PMID 20809437
- [Background] Canadian Medical Association. CMA National Physician Health Survey - A National Snapshot. October 2018.
- [Background] Weng HC, Hung CM, Liu YT, Cheng YJ, Yen CY, Chang CC, Huang CK. Associations between emotional intelligence and doctor burnout, job satisfaction and patient satisfaction. Med Educ. 2011 Aug;45(8):835-42. doi: 10.1111/j.1365-2923.2011.03985.x. PMID 21752080
- [Background] Bianchi R, Schonfeld IS, Laurent E. Burnout-depression overlap: a review. Clin Psychol Rev. 2015 Mar;36:28-41. doi: 10.1016/j.cpr.2015.01.004. Epub 2015 Jan 17. PMID 25638755
- [Background] Dewa CS, Loong D, Bonato S, Thanh NX, Jacobs P. How does burnout affect physician productivity? A systematic literature review. BMC Health Serv Res. 2014 Jul 28;14:325. doi: 10.1186/1472-6963-14-325. PMID 25066375
- [Background] Dewa CS, Jacobs P, Thanh NX, Loong D. An estimate of the cost of burnout on early retirement and reduction in clinical hours of practicing physicians in Canada. BMC Health Serv Res. 2014 Jun 13;14:254. doi: 10.1186/1472-6963-14-254. PMID 24927847
- [Background] Shanafelt TD, Mungo M, Schmitgen J, Storz KA, Reeves D, Hayes SN, Sloan JA, Swensen SJ, Buskirk SJ. Longitudinal Study Evaluating the Association Between Physician Burnout and Changes in Professional Work Effort. Mayo Clin Proc. 2016 Apr;91(4):422-31. doi: 10.1016/j.mayocp.2016.02.001. PMID 27046522
- [Background] Collier R. Physician burnout a major concern. CMAJ. 2017 Oct 2;189(39):E1236-E1237. doi: 10.1503/cmaj.1095496. No abstract available. PMID 28970264
- [Background] Panagioti M, Panagopoulou E, Bower P, Lewith G, Kontopantelis E, Chew-Graham C, Dawson S, van Marwijk H, Geraghty K, Esmail A. Controlled Interventions to Reduce Burnout in Physicians: A Systematic Review and Meta-analysis. JAMA Intern Med. 2017 Feb 1;177(2):195-205. doi: 10.1001/jamainternmed.2016.7674. PMID 27918798
- [Background] Williams ES, Manwell LB, Konrad TR, Linzer M. The relationship of organizational culture, stress, satisfaction, and burnout with physician-reported error and suboptimal patient care: results from the MEMO study. Health Care Manage Rev. 2007 Jul-Sep;32(3):203-12. doi: 10.1097/01.HMR.0000281626.28363.59. PMID 17666991
- [Background] Shanafelt TD, Gorringe G, Menaker R, Storz KA, Reeves D, Buskirk SJ, Sloan JA, Swensen SJ. Impact of organizational leadership on physician burnout and satisfaction. Mayo Clin Proc. 2015 Apr;90(4):432-40. doi: 10.1016/j.mayocp.2015.01.012. Epub 2015 Mar 18. PMID 25796117
- [Background] West CP, Dyrbye LN, Shanafelt TD. Physician burnout: contributors, consequences and solutions. J Intern Med. 2018 Jun;283(6):516-529. doi: 10.1111/joim.12752. Epub 2018 Mar 24. PMID 29505159
- [Derived] Spilg EG, McNeill K, Dodd-Moher M, Dobransky JS, Sabri E, Maniate JM, Gartke KA. Physician Leadership and Its Effect on Physician Burnout and Satisfaction During the COVID-19 Pandemic. J Healthc Leadersh. 2025 Feb 27;17:49-61. doi: 10.2147/JHL.S487849. eCollection 2025. PMID 40034467